CLINICAL TRIAL: NCT00451750
Title: The Efficacy of Cortisol in Combination With Behavioral Therapy in the Treatment of Phobias
Brief Title: Cortisol in the Treatment of Phobias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: University Hospital, Basel, Switzerland (Other)
Responsible Party: Dominique de Quervain, Prof. MD, University of Zurich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007DR3069
Record Dates: First submitted 2007-03-21; First posted 2007-03-23 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Phobia
Keywords: phobia; cortisol; memory; treatment
MeSH Terms: conditions — Phobic Disorders | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Cortisol — 20 mg for 3 times

SUMMARY:
The aim of this prospective, double-blind, placebo-controlled, randomized study is to investigate if glucocorticoid treatment, in combination with exposure therapy, helps to reduce phobic fear in patients with phobia.

ELIGIBILITY:
Inclusion Criteria:

- Female and male patients with a specific phobia (fear of heights) according to DSM-IV criteria.

Exclusion Criteria:

* Severe acute or chronic somatic diseases
* Psychiatric disorder other than specific phobia
* Topic glucocorticoid therapy (for large skin parts)
* Inhaled glucocorticoids
* Psychotropic medication
* Pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
visual analog scales for fear and acrophobia questionnaires | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Dominique JF de Quervain, MD, Prof., Principal Investigator — University of Zurich; Frank Wilhelm, Prof., Principal Investigator — University of Basel
Locations (1):
- University of Basel, Basel, Switzerland

REFERENCES:
- [Background] Soravia LM, Heinrichs M, Aerni A, Maroni C, Schelling G, Ehlert U, Roozendaal B, de Quervain DJ. Glucocorticoids reduce phobic fear in humans. Proc Natl Acad Sci U S A. 2006 Apr 4;103(14):5585-90. doi: 10.1073/pnas.0509184103. Epub 2006 Mar 27. PMID 16567641